CLINICAL TRIAL: NCT01612533
Title: A Registry Study on Safety Surveillance of Shenfu (a Chinese Medicine Injection) Used in China
Brief Title: Safety Study of Shenfu (a Chinese Medicine Injection) Used in Hospitals in China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy Director, China Academy of Chinese Medical Sciences
Other Study IDs: RSCMI-IV
Record Dates: First submitted 2012-06-03; First posted 2012-06-06 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Shock; Coronary Heart Disease
MeSH Terms: conditions — Shock; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study was advocated by Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences in October 2011.

It was funded by China major scientific and technological specialized project for 'significant new formulation of new drugs'.

Shenfu is kind of Chinese Medicine injection used for treating shock and coronary heart disease in many Chinese hospitals.

The purpose of this study is to determine adverse drug events or adverse drug reaction in large sample size 20,000 patients.

DETAILED DESCRIPTION:
Safety surveillance on Chinese Medicine injection is an important problem that needs to be sorted out ,because in mainland China hospitals ,Chinese Medicine Injection are used widely. Population for taking medicine characteristics,the incidence rate of ADR and other uncertain factors influence can not be found now.

A registry study for Shenfu injection safety surveillance with 20000 patients will be conducted from Jan.2012 to Dec.2015.

Eligibility criteria Patients who will use Shenfu injection in selected hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients using Shenfu injection from 2012 to 2014

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An anticipated sample size was caculated in this study, about 20000. Patients using Shenmai injection from 2012 to 2014 in 15 hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events; incidence of Shenfu'ADRs and identify factors that contributed to the occurrence of the adverse reaction. | The registry procedure will last 3 years only for patients using Shenfu.

CONTACTS AND LOCATIONS:
Overall Officials: Yan M Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences